CLINICAL TRIAL: NCT03789175
Title: Exploratory Study of Nicotinamide Riboside on Mitochondrial Function in Li-Fraumeni Syndrome
Brief Title: Nicotinamide Riboside on Mitochondrial Function in Li-Fraumeni Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 190034; 19-H-0034
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2019-11-26

CONDITIONS: Cancer; Skin Fibroblasts; Muscle Weakness
Keywords: Oxidative Phosphorylation Capacity; Increased Oxidative Metabolism; Regeneration of Phosphocreatine (PCr); Inherited Mutation of TP53 Tumor Suppressor Gene
MeSH Terms: conditions — Neoplasms; Muscle Weakness | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nicotinamide riboside (NR) in Li-Fraumeni syndrome (Other): Nicotinamide riboside (NR) to be initiated at week 0 at dose of 250 mg twice a day. At Week 1, NR will be titrated to 500 mg twice a day. At Week 6, NR will be titrated to 750 mg twice a day. At Week 7, NR will be titrated to 1000 mg twice a day or as tolerated until end of week 12. At week 12, if participant responds to primary endpoint, participant will washout of NR at week 18 then restart NR at week 24 until week 30. If there is not response to NR treatment at week 12, the participant may continue taking NR at a tolerated dose until week 24 and the primary endpoint will be re-measured. If participant has a positive response to NR treatment at week 24, then the participant will washout of NR until week 30, at which time the primary endpoint will be re-measured to ensure return to baseline. If there is no response to continued NR treatment at week 24, the study will be ended.
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside (NR) — Niacin is a form of vitamin B3 and has been used to treat hypercholesterolemia for many years. There is growing evidence that nicotinamide adenine dinucleotide (NAD+ can maintain mitochondria through various mechanisms and that it is possible to improve mitochondrial function by dietary supplementation with the vitamin B3 analogue nicotinamide riboside (NR), an intermediate in the NAD+ salvage pathway. We have observed that culturing the fibroblasts of a LFS patient with mitochondrial deficiency in medium containing NR rescues the defect in mitochondrial respiration.
  Other Names: Niagen; Nicotinamide Riboside (NR)

SUMMARY:
Background:

Nicotinamide riboside (NR) is a vitamin B3 dietary supplement. It may help improve muscle function, that may in turn may improve a person s exercise capacity. Researchers want to study how skeletal muscle responds to NR in an individual who has Li-Fraumeni Syndrome and slow muscle energy recovery after exercise.

Objective:

To study how nicotinamide riboside affects skeletal muscle after exercise.

Eligibility:

One person at least 18 years old with Li-Fraumeni syndrome and a certain gene mutation

Design:

The participant will be screened with a medical history, physical exam, and blood and urine tests.

The participant may also have a heart test.

The participant will maintain their regular diet and supplements during the study.

The participant will take the study drug as 1-4 tablets twice a day for 12 weeks. The participant may be contacted with reminders and questions about side effects.

The participant will have 4-5 visits over 18-30 weeks. At visits, the participant will repeat screening tests. At some visits they will also have:

* Ultrasound of the heart with a wand placed on the chest.
* Test of oxygen used at rest and exercise, while wearing a face mask.
* Exercise test on a treadmill or bicycle with electrodes on the skin.
* Magnetic resonance spectroscopy. The participant will have no caffeine for 12 hours. Then they will lie in a machine for about 2 hours. Sometimes they will lie still. Sometimes they will be asked to move.

Health questionnaire

The participant may have a skin sample taken by needle.

The participant will be withdrawn from the study if they become pregnant.

DETAILED DESCRIPTION:
We have previously reported that inherited mutations of TP53, which causes the premature cancer disorder Li-Fraumeni syndrome (LFS), can promote mitochondrial function both in patients and mouse models. In the course of our follow up studies, we encountered a LFS patient with a long-standing history of fatigue and muscle weakness of unclear etiology. Notably, we observed in vivo evidence of markedly decreased mitochondrial function in her leg skeletal muscle during exercise using noninvasive phosphorus-31 magnetic resonance spectroscopy (31P-MRS), a technique that has previously been used to study patients with primary mitochondrial disorders. The decrease in mitochondrial function was also confirmed by the patients skin fibroblasts in vitro using standard biochemical measurements.

There is growing evidence that nicotinamide adenine dinucleotide (NAD+) homeostasis plays a significant role in maintaining the mitochondria through various mechanisms and that it is possible to improve mitochondrial function by dietary supplementation with the vitamin B3 analogue nicotinamide riboside (NR), an intermediate in the NAD+ salvage pathway. Remarkably, we observed that culturing the LFS patients fibroblasts in medium containing NR rescued the severe deficit in mitochondrial respiration. While continuing our investigations into the molecular mechanism(s) underlying the mitochondrial dysfunction observed in this patient, the in vitro rescue of the respiratory deficiency by NR presents a unique opportunity to investigate whether it can also be observed in vivo using skeletal muscle 31P-MRS. We propose to explore the effect of NR, currently available as a dietary supplement, on in vivo mitochondrial function in this LFS patient.

ELIGIBILITY:
* INCLUSION CRITERIA:
* At least 18-years of age and able to give informed consent
* Have delayed phosphocreatine (PCr) recovery time constant >45 sec by 31P-magnetic resonance spectroscopy (MRS) testing and a history of fatigue symptoms
* Ability to undergo study procedures, including scheduled visits, blood draws and skeletal muscle exercise Nuclear Magnetic Resonance (NMR)
* Have Li-Fraumeni syndrome and confirmed TP53 mutation by genetic testing
* Committed to using reliable contraception which may include abstinence during study participation
* Female participants of child-bearing ability and potential willing to commit to reliable contraception while participating in the study

EXCLUSION CRITERIA:

* Current systemic treatment for cancer
* Unable to perform required study visits or procedures
* Magnetic resonance imaging (MRI) incompatible hardware
* Pregnant or breastfeeding women
* History of intolerance to NR precursor compounds, including niacin or nicotinamide

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Hwang, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-H-0034.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a one-subject study so there are no recruitment or screening of other subjects.
Period: Week 0 to Week 12 of NR
Arm/Group | Nicotinamide Riboside (NR) in Li-Fraumeni Syndrome
Started | 1
Completed | 1
Not Completed | 0
Period: Week 12 to Week 24 of NR
Arm/Group | Nicotinamide Riboside (NR) in Li-Fraumeni Syndrome
Started | 1
Completed | 1 (Participant did not meet primary endpoint and completed study at week 24)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nicotinamide Riboside (NR) in Li-Fraumeni Syndrome
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in PCr Recovery Tc Measurement From Baseline to 12 Week NR Supplementation Using the 31P-MRS Skeletal Muscle Submaximal Exercise.
Description: The effect of nicotinamide riboside (NR) supplementation on the phosphocreatine (PCr) recovery time constant (Tc) of skeletal muscle after exercise as a marker of mitochondrial oxidative phosphorylation capacity.
  The phosphocreatine level will be measured using 31P-magnetic resonance spectroscopy (MRS) during the following sequence of 3-minute rest, 2-minute exercise, and 6-minute recovery periods. The 31P spectra will be obtained during these periods and analyzed with the use of SAGE 7 (GE Healthcare) and IDL, version 6.4 (Exelis Visual Information Solutions), software. The single exponential recovery time constant (Tc) is calculated from the post-exercise recovery period data.
Time Frame: Baseline to 12 weeks
Measure: Number; unit: Seconds
Groups:
- Baseline Phosphocreatine (PCr) Recovery Tc Measurement: All participants prior to initiation of nicotinamide riboside (NR).
Arm/Group | Baseline Phosphocreatine (PCr) Recovery Tc Measurement | Nicotinamide Riboside (NR) in Li-Fraumeni Syndrome
Number analyzed (Participants) | 1 | 1
Seconds | 60 | 73

2. Secondary Outcome: Change in Time of CPET Time as a Measure of Exercise Tolerance From Baseline to 12 Weeks of NR Supplementation.
Description: Measure change in time of cardiopulmonary exercise test (CPET) to determine exercise tolerance from baseline to 12 weeks of NR supplementation.
Time Frame: Baseline to 12 weeks
Measure: Number; unit: Minutes
Groups:
- Baseline CPET Exercise Endurance Time: All participants prior to initiation of nicotinamide riboside (NR).
Arm/Group | Baseline CPET Exercise Endurance Time | Nicotinamide Riboside (NR) in Li-Fraumeni Syndrome
Number analyzed (Participants) | 1 | 1
Minutes | 12.1 | 11.68

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Nicotinamide Riboside (NR) in Li-Fraumeni Syndrome
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotinamide Riboside (NR) in Li-Fraumeni Syndrome (N=1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Metabolism and nutrition disorders) | 1 (1)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT03789175/Prot_SAP_000.pdf